CLINICAL TRIAL: NCT05818891
Title: Prospective, Multicenter, Non-Controlled, Non-Randomized, Open-Label Study To Evaluate The Efficacy And Performance Of The Mpact® Dual Mobility Hemispheric Cup
Brief Title: Multicenter Mpact DM France
Status: Recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P01.017.03
Record Dates: First submitted 2023-04-05; First posted 2023-04-19 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Total Hip Arthroplasty; Survival, Prosthesis
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary objective of the study is to evaluate the 10-year performance of the MPACT DM cup in the treatment of patients requiring total hip arthroplasty.

The primary endpoint is the 10-year life span of the prosthesis according to the Kaplan Meier curve.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the 10-year performance of the MPACT DM cup in the treatment of patients requiring total hip arthroplasty evaluated through the Kaplan Meier curve.

The secondary objectives of the study are:

* To assess the function of the operated hip
* Evaluate the safety of the implant
* Evaluate the stability of the prosthetic components

Secondary endpoints were:

* Harris Hip Score The Harris Hip Score (HHS) items include an analysis of the operated hip according to pain, function, mobility and stability and a deformity analysis. The Harris Hip Score will be used to assess the patient's subjective and objective improvement in the above criteria.
* Evaluation of standard radiographs from the front and side. Periprosthetic edging and osteolysis will be evaluated using Delee and Charnley zones for the acetabular component and Gruen zones for the femoral component.
* Evaluation of implant stability and fit using the ARA score. This score is used to determine whether the implant causes changes in the surrounding bone structures. If signs occur, they can be considered either as "neutral", showing a simple adaptation and not reducing the result, or as "negative" to varying degrees. The maximum ARA score is 6 points, negative points from 1 to 4 can be attributed for each of these "negative" signs.

The arithmetic summation of these "risk factors" will lead to a final "score", defining the adaptation of the prosthesis to the bone sleeve at the time the images are taken, and which may naturally vary with time, either positively, if the fixation, which was precarious at the time, stabilizes (secondary osteoinduction by Hydroxyapatite of initial fibrosis zones, for example), or negatively in the presence of an evolving destabilization (there is obviously no negative score). The approach is similar for the femur and for the acetabulum.

❖ Collection of intraoperative and postoperative complications. Complications, such as infection, loosening, deep vein thrombosis (DVT), fracture, as well as other unexpected complications, will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a disease that meets the indications for use of Medacta implants (according to the instructions for use)
2. Patient eligible for first-line total hip replacement
3. Patient between 18 and 80 years of age
4. Patient covered by the Social Security system or an equivalent protection plan
5. Patient who is capable, in the opinion of the investigator, of fulfilling the requirements of the study

Exclusion Criteria:

1. Patient requiring a transplant
2. Patient with progressive local or systemic infection
3. Patient with muscle loss, neuromuscular disease, or vascular impairment of the affected limb making surgery unwarranted
4. Patient with known medical problems that may compromise independent recovery of mobility
5. Patient with a BMI greater than 40 kg/m².
6. Patient with major cognitive problems that do not allow a good understanding of the study requirements
7. Patient living in a geographical area that does not allow the study follow-up
8. Patient participating in interventional research.
9. Minor patient
10. Protected adult patient
11. Vulnerable person according to article L1121-6 of the Public Health Code
12. Pregnant or nursing woman.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The total number of patients needed for this study is 600. All patients with a condition requiring hip joint replacement will be invited to participate in the study by the investigator during consultations.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-04-05 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate the 10-year performance of the MPACT DM cup in the treatment of patients requiring total hip arthroplasty. | 10 years after the index surgery
  Analysis with Kaplan Meier curve considering the revisions of the implants

SECONDARY OUTCOMES:
Evaluate the function of the operated hip | pre-op, 3 months, 1 year, 3 years, 5 years and 10 years after the index surgery
  Evaluation of the Harris Hip Score with the analysis of the operated hip for pain, function, mobility and stability and a deformity analysis.
  The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. Results can be recorded and calculated online. The maximum score possible is 100. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent
  Evaluation of standard radiographs from the front and side. Periprosthetic edging and osteolysis will be evaluated using Delee and Charnley zones for the acetabular component and Gruen zones for the femoral component.
To evaluate the safety of the implant | Intra-op, 3 months, 1 year, 3 years, 5 years and 10 years after the index surgery
  Collecting all the adverse events through time
  Collection of intraoperative and postoperative complications. Complications, such as infection, loosening, deep vein thrombosis (DVT), fracture, as well as other unexpected complications, will be evaluated.
To evaluate the stability of the prosthetic components | pre-op, 3 months, 1 year, 3 years, 5 years and 10 years after the index surgery
  Evaluation of implant stability and fit using the ARA score. This score is used to determine whether the implant causes changes in the surrounding bone structures. If signs occur, they can be considered either as "neutral", showing a simple adaptation and not reducing the result, or as "negative" to varying degrees. The maximum ARA score is 6 points, negative points from 1 to 4 can be attributed for each of these "negative" signs.
  The arithmetic summation of these "risk factors" will lead to a final "score", defining the adaptation of the prosthesis to the bone sleeve at the time the images are taken, and which may naturally vary with time, either positively, if the fixation, which was precarious at the time, stabilizes (secondary osteoinduction by Hydroxyapatite of initial fibrosis zones, for example), or negatively in the presence of an evolving destabilization (there is obviously no negative score). The approach is similar for the femur and for the acetabulum.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DEROCHE, Principal Investigator — Centre Orthopédique Médico-Chirurgical de Dracy Le Fort
Locations (1):
- Centre Orthopédique Médico-Chirurgical de Dracy Le Fort, Dracy-le-Fort, France

IPD SHARING:
Plan to Share IPD: No